CLINICAL TRIAL: NCT06755879
Title: the Impact of a Digital Game-based Learning Activity on Nursing Students' Learning and Motivation Levels Regarding Surgical Site Infection Prevention Initiatives
Brief Title: the Impact of a Digital Game-based Learning Activity on Nursing Students' Understanding of Surgical Site Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Collaborators: University of Gaziantep (Other)
Responsible Party: Principal Investigator, hatice akaltun, Lecturer, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VYYU-SBF-HAKALTUN-001
Record Dates: First submitted 2024-12-18; First posted 2025-01-01 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Surgical Site Infections; Education
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- digital game-based learning activity group (Experimental): the level of learning interventions to prevent surgical site infections with digital game-based learning activity will be evaluated with pre-test and post-test
  Interventions: Behavioral: digital game-based learning activity
- theoretical course group (Active Comparator): the level of learning the theoretical course and interventions to prevent surgical site infections will be evaluated with pre-test and post-test
  Interventions: Behavioral: traditional method
- control group (No Intervention): The control group will be evaluated only with the pre-test post-test without any intervention.

INTERVENTIONS:
Behavioral: digital game-based learning activity — learning interventions to prevent surgical site infections with a digital game-based learning activity
  Arms: digital game-based learning activity group
Behavioral: traditional method — Evaluation of the effectiveness of students' learning of interventions to prevent surgical site infections in the theoretical course taught by traditional method
  Arms: theoretical course group

SUMMARY:
The aim of this randomized controlled trial was to evaluate the effect of a digital game-based learning activity on students' learning of interventions to prevent surgical site infections.This study will seek answers to the following questions:

Is digital game-based learning activity effective in students' learning process? Is the traditional method of theoretical lecturing effective in the learning process? What is the effect of students' learning methods on their motivation? The researchers will compare the group with the theoretical lecture to see the effectiveness of the digital game-based learning activity.

Participants will be divided into 3 groups. In the first group, the level of learning interventions to prevent surgical site infections with digital game-based learning activity will be evaluated with pre-test and post-test In the second group, the level of learning the theoretical course and interventions to prevent surgical site infections will be evaluated with pre-test and post-test.

The control group will be evaluated only with the pre-test post-test without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Having a cell phone, computer or tablet device.

  * To have internet access on one of the cell phone, computer or tablet devices.
  * To have taken the Surgical Diseases Nursing course.
  * To be a 4th year student of Van Yüzüncü Yıl University Faculty of Health Sciences, Department of Nursing
  * Volunteering to participate in the research

Exclusion Criteria:

* - Graduating from a health vocational high school or coming from a health-related department with vertical transfer
* Limited ability to read and write in Turkish.
* Not having a software infrastructure suitable for opening digital game activities on mobile phones, computers or tablet devices

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
pre-test post-test question form | after the pre-test is applied, the digital game-based learning activity will be used for 5 days. the post-test will be applied 3 weeks after the pre-test
  the effectiveness of the digital game-based learning activity will be measured by pre-test post-test (Measurement will be made with a pre-test post-test prepared by the researcher.)

SECONDARY OUTCOMES:
pre-test post-test question form | After the pre-test is applied, a 45-minute theoretical lesson will be held with the students. Post-test will be applied 3 weeks after the pre-test
  pre-test post-test will be applied to evaluate the effectiveness of theoretical explanation with traditional method (Measurement will be made with a pre-test post-test prepared by the researcher.)

OTHER OUTCOMES:
the effect of teaching methods on student motivation | measurement will be made with 3 weeks between pre-test and post-test
  'Teaching material motivation scale' will be applied at the end of the study to determine the effect of teaching methods on student motivation This scale is used to determine the motivation towards a material based on a single application where the user is only dependent on the material. A high score on the total or average score of the scale indicates that the individual's motivation towards the material being evaluated is positively high.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl Üniversitesi /Sağlık Bilimleri Fakültesi, Van, Turkey (Türkiye)